CLINICAL TRIAL: NCT01934140
Title: A PHASE IIIB, OPEN, MULTI-CENTER STUDY TO EVALUATE THE LONG-TERM ANTIBODY PERSISTENCE AT 6, 7, 8, 9 AND 10 YEARS AFTER THE ADMINISTRATION OF ONE DOSE OF MENINGOCOCCAL CONJUGATE VACCINE MENACWY-TT VERSUS ONE DOSE OF MENINGOCOCCAL POLYSACCHARIDE VACCINE MENCEVAX(REGISTERED) ACWY, AND TO EVALUATE THE SAFETY AND IMMUNOGENICITY OF A BOOSTER DOSE OF MENACWY-TT VACCINE ADMINISTERED 10 YEARS AFTER PRIMARY VACCINATION OF 11-55 YEAR OLD SUBJECTS WITH MENACWY-TT OR MENCEVAX (REGISTERED) ACWY.
Brief Title: Study to Evaluate the Long-term Antibody Persistence of GlaxoSmithKline (GSK) Biologicals' MenACWY-TT Vaccine (GSK134612) Versus Mencevax ACWY in Healthy Adolescents and Adults and Booster Response to MenACWY-TT Vaccine Administered at 10 Years Post-primary Vaccination
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MENACWY-TT-099; 2012-005639-10 (EudraCT Number); C0921002 (Other: Alias Study Number); 116725 (Other: Alias Study Number)
Record Dates: First submitted 2013-08-22; First posted 2013-09-04 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-07

CONDITIONS: Infections, Meningococcal
Keywords: Healthy; Adults; Safety; Neisseria meningitidis; Booster response; Immunogenicity; Adolescents; Serogroups A, C, W-135, and Y; long-term antibody persistence
MeSH Terms: conditions — Meningococcal Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACWY-TT group (Experimental): All subjects vaccinated with MenACWY-TT in study MENACWY-TT-015 will be assigned to this group. At Month 120 after primary vaccination, these subjects will be vaccinated with a booster dose of MenACWY-TT in this study.
  Interventions: Biological: Meningococcal vaccine GSK134612
- MenPS group (Active Comparator): All subjects vaccinated with Mencevax ACWY in study MENACWY-TT-015 will be assigned to this group. At Month 120 after primary vaccination, these subjects will be vaccinated with a dose of MenACWY-TT in this study.
  Interventions: Biological: Meningococcal vaccine GSK134612

INTERVENTIONS:
Biological: Meningococcal vaccine GSK134612 — 1 dose administered intramuscularly in the non-dominant deltoid region.

SUMMARY:
The purpose of this study is to evaluate the long-term antibody persistence from 6, 7, 8, 9 to 10 years post-administration of MenACWY-TT conjugate vaccine as compared to Mencevax ACWY when given to healthy subjects 11 to 55 years of age. In addition, the safety and immunogenicity of a booster dose of MenACWY-TT vaccine administered to all eligible subjects 10 years after the primary vaccination will be evaluated.

All Filipino subjects who received the primary vaccination in the primary vaccination study 107386 (NCT00356369) will be invited to enrol in the long-term follow up and booster phase. No new subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy the following criteria at study entry to the persistence phase:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol. Or /and subjects' parent(s)/Legally Acceptable Representative(s) [LAR(s)] who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* A male or female between and including 17 and 66 years of age at the time of entry into the present study.
* Has completed the vaccination phase of the vaccination study MENACWY-TT-015.
* In alignment with local laws and regulations, written informed consent obtained from parents/LAR(s) of the subject and written informed assent obtained from the subject if the subject is less than 18 years of age, or written informed consent obtained from the subject if the subject has achieved the 18th birthday. The subjects ≥18 years of age at the time of enrollment will sign the informed consent form, even if the parent/ LAR previously signed the ICF before the subject reached the legal age of consent.
* Healthy subjects as established by medical history and history-directed physical examination before entering into the study.

All subjects must satisfy the following additional criteria prior to entry of the booster phase:

* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Child in care.
* Previous vaccination with meningococcal polysaccharide or conjugate vaccine outside of study MENACWY-TT-015.
* History of meningococcal disease due to serogroup A, C, W-135 or Y.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including Human Immunodeficiency Virus (HIV) infection, based on medical history and physical examination.
* Major congenital defects or serious chronic illness.
* Family history of congenital or hereditary immunodeficiency.
* History of chronic alcohol consumption and/or drug abuse.

Additional exclusion criteria for booster phase at Month 120 study entry (to be checked at Month 120) for all subjects

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the booster dose of study vaccine, or planned use during the follow-up period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs within six months prior to the booster vaccine dose. Inhaled and topical steroids are allowed.
* Administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the booster dose of study vaccine or planned administration within 30 days after vaccination (with the day of vaccination considered Day 0), with the exception of a licensed inactivated influenza vaccine.
* Administration of immunoglobulins and/or any blood products within the three months preceding the booster vaccination or planned administration during the follow-up period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Previous vaccination with tetanus toxoids within the last month.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* History of any neurological disorders or seizures, including Guillain-Barré syndrome (GBS). History of a simple, single febrile seizure is permitted.
* Acute disease and/or fever at the time of enrollment.

  * Fever is defined as temperature ≥ 37.5°C for oral, axillary or tympanic route, or ≥ 38.0°C for rectal route. The preferred route for recording temperature in this study will be oral.
  * Subjects with a minor illness without fever may, be enrolled at the discretion of the investigator.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Ages: 17 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Philippines (2):
  - Research Institute for Tropical Medicine, Muntinlupa City, National Capital Region
  - Philippine General Hospital, Manila

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Borja-Tabora CFC, Peyrani P, Webber C, Van der Wielen M, Cheuvart B, De Schrevel N, Bianco V, Aris E, Cutler M, Li P, Perez JL. A phase 2b/3b MenACWY-TT study of long-term antibody persistence after primary vaccination and immunogenicity and safety of a booster dose in individuals aged 11 through 55 years. BMC Infect Dis. 2020 Jun 18;20(1):426. doi: 10.1186/s12879-020-05104-5. PMID 32552685
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=MENACWY-TT-099&StudyName=A+Phase+Iiib%2C+Open%2C+Multi-center+Study+To+Evaluate+The+Long-term+Antibody+Persistence+At+6%2C+7%2C+8%2C+9+And+10+Years+After+The+Administration+Of+One+Dose+Of+Meningococcal+Conjugate+Vaccine+Menacwy-tt+Versus+One+Dose+Of+Meningococcal+Polysaccharide+Vaccine+Mencevax%28registered%29+Acwy%2C+And+To+Evaluate+The+Safety+And+Immunogenicity+Of+A+Booster+Dose+Of+Menacwy-tt+Vaccine+Administered+10+Years+After+Primary+Vaccination+Of+11-55+Year+Old+Subjects+With+Menacwy-tt+Or+Mencevax+%28registered%29+Acwy.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment for this study (MENACWY-TT-99) started at Year 6 post primary vaccination in study 107386 [NCT00356369]. However, as approval was not obtained from authorities until after end of Year 6, hence no planned activities was done for Year 6.
Pre-assignment Details: In this study, participants from the study 107386 [NCT00356369] were followed up for assessment of persistence of immune response. And those who consented received booster vaccination and were followed up for another 6 months.
Groups:
- ACWY-TT Group: Persistence phase was followed up by booster phase. Persistence phase: Participants received a single 0.5 millilitre (mL) dose of meningococcal serogroups A, C, W-135, Y tetanus toxoid conjugate (MenACWY-TT) vaccine intramuscularly, as primary vaccination in study 107386 [NCT00356369]. Then, in this study (MENACWY-TT-99), they were evaluated for long-term persistence of immune response for 4 years (7, 8, 9 and 10 years post primary vaccination). Booster phase: All eligible participants from persistence phase who provided informed consent to enroll in booster phase, received a single 0.5 mL booster dose of MenACWY-TT vaccine intramuscularly in this study, 10 years post primary vaccination in 107386 [NCT00356369], and were followed up for 6 months after booster vaccination.
- MenPS Group: Persistence phase was followed up by booster phase. Persistence phase: Participants received a single 0.5 mL dose of Mencevax ACWY vaccine intramuscularly, as primary vaccination in study 107386 [NCT00356369]. Then, in this study (MENACWY-TT-99) they were evaluated for long-term persistence of immune response for 4 years (7, 8, 9 and 10 years post primary vaccination). Booster phase: All eligible participants from persistence phase who provided informed consent to enroll in booster phase, received a single 0.5 mL booster dose of MenACWY-TT vaccine intramuscularly in this study, 10 years post primary vaccination, and were followed up for 6 months after booster vaccination.
Period: Persistence Phase (Year 6-10)
Arm/Group | ACWY-TT Group | MenPS Group
Started | 235 | 76
Completed | 152 (Participants completed all persistence phase visits) | 51 (Participants completed all persistence phase visits)
Not Completed | 83 | 25
Not completed — Other | 24 | 6
Not completed — Lost to Follow-up | 5 | 2
Not completed — Migrated/moved from study area | 31 | 10
Not completed — Eligibility criteria not fulfilled | 2 | 0
Not completed — Missed at least 1 persistence visit | 21 | 7
Period: Booster Phase (6 Months)
Arm/Group | ACWY-TT Group | MenPS Group
Started | 164 (Eligible participants from persistence phase who provided consent, were enrolled in booster phase.) | 56 (Eligible participants from persistence phase who provided consent, were enrolled in booster phase.)
Vaccinated | 164 | 56
Completed | 159 | 53
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Missed at least 1 booster visit | 2 | 1
Not completed — Migrated/moved from study area | 2 | 2

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all the participants enrolled in the study.
Groups:
- ACWY-TT Group: Persistence phase was followed up by booster phase. Persistence phase: Participants received a single 0.5 mL dose of MenACWY-TT vaccine intramuscularly, as primary vaccination in study 107386 [NCT00356369]. Then, in this study (MENACWY-TT-99), they were evaluated for long-term persistence of immune response for 4 years (7, 8, 9 and 10 years post primary vaccination). Booster phase: All eligible participants from persistence phase who provided informed consent to enroll in booster phase, received a single 0.5 mL booster dose of MenACWY-TT vaccine intramuscularly in this study, 10 years post primary vaccination in 107386 [NCT00356369], and were followed up for 6 months after booster vaccination.
- Total: Total of all reporting groups
Arm/Group | ACWY-TT Group | MenPS Group | Total
Number analyzed (Participants) | 235 | 76 | 311
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (8.2) | 25.2 (8.4) | 25.2 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 40 | 148
  Male | 127 | 36 | 163
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 235 | 76 | 311
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 235 | 76 | 311
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Persistence Phase: Percentage of Participants With Serum Bactericidal Assay Using Rabbit Complement (rSBA) Titers Greater Than or Equal to (>=) 1:8 and >=1:128 For Each of the 4 Serogroups After 6 Years of Primary Vaccination
Description: Serogroups included neisseria meningitidis serogroup A (MenA), Neisseria meningitidis serogroup C (MenC), Neisseria meningitidis serogroup W-135 (MenW-135) and Neisseria meningitidis serogroup Y (MenY).
Time Frame: After 6 years of primary vaccination
Population: Data was not collected and analyzed for this outcome measure because approval was not obtained from the authorities for Year 6 activities.
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Persistence Phase: Percentage of Participants With rSBA Titers >= 1:8 and >=1:128 For Each of the 4 Serogroups After 7 Years of Primary Vaccination
Description: Serogroups included MenA, MenC, MenW-135 and MenY.
Time Frame: After 7 years of primary vaccination
Population: All eligible participants who received primary vaccination with MenACWY-TT or Mencevax ACWY during study 107386 [NCT00356369], had available assay results for at least 1 tested antigen. Here, "Overall Number of Participants Analyzed" (N) signifies number of participants evaluable for this measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 206 | 65
percentage of participants
  rSBA-MenA: >=1:8 | 88.3 [83.2 to 92.4] | 67.7 [54.9 to 78.8]
  rSBA-MenC: >=1:8 | 82.5 [76.6 to 87.4] | 76.9 [64.8 to 86.5]
  rSBA-MenW-135: >=1:8 | 60.7 [53.7 to 67.4] | 23.1 [13.5 to 35.2]
  rSBA-MenY: >=1:8 | 80.1 [74.0 to 85.3] | 46.2 [33.7 to 59.0]
  rSBA-MenA: >=1:128 | 73.8 [67.2 to 79.7] | 46.2 [33.7 to 59.0]
  rSBA-MenC: >=1:128 | 61.7 [54.6 to 68.3] | 61.5 [48.6 to 73.3]
  rSBA-MenW-135: >=1:128 | 52.4 [45.4 to 59.4] | 16.9 [8.8 to 28.3]
  rSBA-MenY: >=1:128 | 76.7 [70.3 to 82.3] | 38.5 [26.7 to 51.4]

3. Primary Outcome: Persistence Phase: Percentage of Participants With rSBA Titers >= 1:8 and >=1:128 For Each of the 4 Serogroups After 8 Years of Primary Vaccination
Description: Serogroups included MenA, MenC, MenW-135 and MenY.
Time Frame: After 8 years of primary vaccination
Population: All eligible participants who received primary vaccination with MenACWY-TT or Mencevax ACWY during study 107386 [NCT00356369], had available assay results for at least 1 tested antigen. Here, "N" signifies number of participants evaluable for this measure and "Number analyzed" (n): participants analyzed for specified serogroup.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 208 | 67
percentage of participants
  rSBA-MenA: >=1:8 | 76.0 [69.6 to 81.6] | 56.7 [44.0 to 68.8]
  rSBA-MenC: >=1:8: number analyzed (Participants) | 204 | 67
  rSBA-MenC: >=1:8 | 86.3 [80.8 to 90.7] | 80.6 [69.1 to 89.2]
  rSBA-MenW-135: >=1:8: number analyzed (Participants) | 207 | 67
  rSBA-MenW-135: >=1:8 | 66.2 [59.3 to 72.6] | 23.9 [14.3 to 35.9]
  rSBA-MenY: >=1:8: number analyzed (Participants) | 206 | 67
  rSBA-MenY: >=1:8 | 76.2 [69.8 to 81.9] | 40.3 [28.5 to 53.0]
  rSBA-MenA: >=1:128 | 60.6 [53.6 to 67.3] | 40.3 [28.5 to 53.0]
  rSBA-MenC: >=1:128: number analyzed (Participants) | 204 | 67
  rSBA-MenC: >=1:128 | 68.1 [61.3 to 74.5] | 64.2 [51.5 to 75.5]
  rSBA-MenW-135: >=1:128: number analyzed (Participants) | 207 | 67
  rSBA-MenW-135: >=1:128 | 60.9 [53.9 to 67.6] | 16.4 [8.5 to 27.5]
  rSBA-MenY: >=1:128: number analyzed (Participants) | 206 | 67
  rSBA-MenY: >=1:128 | 70.9 [64.2 to 77.0] | 37.3 [25.8 to 50.0]

4. Primary Outcome: Persistence Phase: Percentage of Participants With rSBA Titers >= 1:8 and >=1:128 For Each of the 4 Serogroups After 9 Years of Primary Vaccination
Description: Serogroups included MenA, MenC, MenW-135 and MenY.
Time Frame: After 9 years of primary vaccination
Population: All eligible participants who received primary vaccination with MenACWY-TT or Mencevax ACWY during study 107386 [NCT00356369], had available assay results for at least 1 tested antigen. Here, "N" signifies number of participants evaluable for this measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 190 | 61
percentage of participants
  rSBA-MenA: >=1:8 | 82.6 [76.5 to 87.7] | 65.6 [52.3 to 77.3]
  rSBA-MenC: >=1:8 | 89.5 [84.2 to 93.5] | 90.2 [79.8 to 96.3]
  rSBA-MenW-135: >=1:8 | 55.8 [48.4 to 63.0] | 9.8 [3.7 to 20.2]
  rSBA-MenY: >=1:8 | 89.5 [84.2 to 93.5] | 57.4 [44.1 to 70.0]
  rSBA-MenA: >=1:128 | 75.3 [68.5 to 81.2] | 59.0 [45.7 to 71.4]
  rSBA-MenC: >=1:128 | 66.8 [59.7 to 73.5] | 67.2 [54.0 to 78.7]
  rSBA-MenW-135: >=1:128 | 50.5 [43.2 to 57.8] | 9.8 [3.7 to 20.2]
  rSBA-MenY: >=1:128 | 86.3 [80.6 to 90.9] | 50.8 [37.7 to 63.9]

5. Primary Outcome: Persistence Phase: Percentage of Participants With rSBA Titers >= 1:8 and >=1:128 For Each of the 4 Serogroups After 10 Years of Primary Vaccination
Description: Serogroups included MenA, MenC, MenW-135 and MenY.
Time Frame: After 10 years of primary vaccination
Population: All eligible participants who received primary vaccination with MenACWY-TT or Mencevax ACWY during study 107386 [NCT00356369], had available assay results for at least 1 tested antigen. Here, "N" signifies number of participants evaluable for this measure and "n": participants analyzed for specified serogroup.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 162 | 54
percentage of participants
  rSBA-MenA: >=1:8 | 76.5 [69.3 to 82.8] | 70.4 [56.4 to 82.0]
  rSBA-MenC: >=1:8: number analyzed (Participants) | 161 | 54
  rSBA-MenC: >=1:8 | 90.7 [85.1 to 94.7] | 88.9 [77.4 to 95.8]
  rSBA-MenW-135: >=1:8: number analyzed (Participants) | 161 | 54
  rSBA-MenW-135: >=1:8 | 70.2 [62.5 to 77.1] | 24.1 [13.5 to 37.6]
  rSBA-MenY: >=1:8: number analyzed (Participants) | 161 | 54
  rSBA-MenY: >=1:8 | 87.0 [80.8 to 91.7] | 64.8 [50.6 to 77.3]
  rSBA-MenA: >=1:128 | 67.9 [60.1 to 75.0] | 57.4 [43.2 to 70.8]
  rSBA-MenC: >=1:128: number analyzed (Participants) | 161 | 54
  rSBA-MenC: >=1:128 | 72.7 [65.1 to 79.4] | 68.5 [54.4 to 80.5]
  rSBA-MenW-135: >=1:128: number analyzed (Participants) | 161 | 54
  rSBA-MenW-135: >=1:128 | 64.6 [56.7 to 72.0] | 22.2 [12.0 to 35.6]
  rSBA-MenY: >=1:128: number analyzed (Participants) | 161 | 54
  rSBA-MenY: >=1:128 | 83.2 [76.5 to 88.6] | 53.7 [39.6 to 67.4]

6. Primary Outcome: Persistence Phase: Geometric Mean Titers With rSBA for Each of the 4 Serogroups After 6 Years of Primary Vaccination
Description: Serogroups included MenA, MenC, MenW-135 and MenY. rSBA titers expressed as the reciprocal of the highest serum last dilution resulting in at least 50 percentage (%) reduction of meningococcal colony-forming units.
Time Frame: After 6 years of primary vaccination
Population: as for outcome 1
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Persistence Phase: Geometric Mean Titers With rSBA for Each of the 4 Serogroups After 7 Years of Primary Vaccination
Description: Serogroups included MenA, MenC, MenW-135 and MenY. rSBA titers expressed as the reciprocal of the highest serum last dilution resulting in at least 50 % reduction of meningococcal colony-forming units.
Time Frame: After 7 years of primary vaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 206 | 65
titers
  rSBA-MenA | 220.8 [167.2 to 291.5] | 54.5 [31.1 to 95.8]
  rSBA-MenC | 105.3 [79.7 to 139.1] | 156.7 [82.7 to 297.1]
  rSBA-MenW-135 | 83.2 [57.0 to 121.5] | 10.0 [6.3 to 15.9]
  rSBA-MenY | 270.2 [195.2 to 373.8] | 32.7 [17.8 to 60.1]

8. Primary Outcome: Persistence Phase: Geometric Mean Titers With rSBA for Each of the 4 Serogroups After 8 Years of Primary Vaccination
Description: as for outcome 7
Time Frame: After 8 years of primary vaccination
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 208 | 67
titers
  rSBA-MenA | 104.8 [77.1 to 142.4] | 44.1 [24.3 to 80.0]
  rSBA-MenC: number analyzed (Participants) | 204 | 67
  rSBA-MenC | 155.4 [118.3 to 204.0] | 240.6 [125.4 to 461.8]
  rSBA-MenW-135: number analyzed (Participants) | 207 | 67
  rSBA-MenW-135 | 119.7 [82.8 to 173.1] | 10.8 [6.7 to 17.5]
  rSBA-MenY: number analyzed (Participants) | 206 | 67
  rSBA-MenY | 181.6 [130.2 to 253.3] | 26.0 [14.5 to 46.6]

9. Primary Outcome: Persistence Phase: Geometric Mean Titers With rSBA for Each of the 4 Serogroups After 9 Years of Primary Vaccination
Description: as for outcome 7
Time Frame: After 9 years of primary vaccination
Population: All eligible participants who received primary vaccination with MenACWY-TT or Mencevax ACWY during study 107386 [NCT00356369], had available assay results for at least 1 tested antigen.Here, "N" signifies number of participants evaluable for this measure.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 190 | 61
titers
  rSBA-MenA | 227.8 [165.0 to 314.5] | 81.2 [44.2 to 149.4]
  rSBA-MenC | 173.3 [129.9 to 231.1] | 264.9 [147.7 to 474.9]
  rSBA-MenW-135 | 71.7 [48.0 to 107.0] | 6.7 [4.5 to 10.0]
  rSBA-MenY | 460.6 [346.2 to 612.7] | 57.8 [30.6 to 109.2]

10. Primary Outcome: Persistence Phase: Geometric Mean Titers With rSBA for Each of the 4 Serogroups After 10 Years of Primary Vaccination
Description: as for outcome 7
Time Frame: After 10 years of primary vaccination
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 162 | 54
titers
  rSBA-MenA | 142.5 [100.4 to 202.1] | 73.7 [40.9 to 132.8]
  rSBA-MenC: number analyzed (Participants) | 161 | 54
  rSBA-MenC | 181.4 [134.6 to 244.4] | 234.0 [122.3 to 447.9]
  rSBA-MenW-135: number analyzed (Participants) | 161 | 54
  rSBA-MenW-135 | 161.5 [104.8 to 248.9] | 11.9 [6.8 to 21.0]
  rSBA-MenY: number analyzed (Participants) | 161 | 54
  rSBA-MenY | 387.0 [274.1 to 546.4] | 63.2 [33.4 to 119.6]

11. Secondary Outcome: Booster Phase: Percentage of Participants With rSBA Titers >=1:8 and >=1:128 For Each of the 4 Serogroups at 1 Month After Booster Vaccination
Description: Serogroups included MenA, MenC, MenW-135 and MenY.
Time Frame: 1 month after booster vaccination
Population: All eligible participants who received primary vaccination in study107386 [NCT00356369], received booster dose of vaccine in study MENACWY-099; for whom assay results are available for antibodies against at least 1 study vaccine antigen component for blood sample taken 1 month after vaccination. N=number of participants evaluable for this measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 155 | 52
percentage of participants
  rSBA-MenA: >=1:8 | 100.0 [97.6 to 100.0] | 100.0 [93.2 to 100.0]
  rSBA-MenC: >=1:8 | 100.0 [97.6 to 100.0] | 98.1 [89.7 to 100.0]
  rSBA-MenW-135: >=1:8 | 100.0 [97.6 to 100.0] | 98.1 [89.7 to 100.0]
  rSBA-MenY: >=1:8 | 100.0 [97.6 to 100.0] | 100.0 [93.2 to 100.0]
  rSBA-MenA: >=1:128 | 100.0 [97.6 to 100.0] | 100.0 [93.2 to 100.0]
  rSBA-MenC: >=1:128 | 100.0 [97.6 to 100.0] | 96.2 [86.8 to 99.5]
  rSBA-MenW-135: >=1:128 | 100.0 [97.6 to 100.0] | 98.1 [89.7 to 100.0]
  rSBA-MenY: >=1:128 | 100.0 [97.6 to 100.0] | 100.0 [93.2 to 100.0]

12. Secondary Outcome: Booster Phase: Geometric Mean Titers With rSBA for Each of the 4 Serogroups at 1 Month After Booster Vaccination
Description: as for outcome 7
Time Frame: 1 month after booster vaccination
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 155 | 52
titers
  rSBA-MenA | 4059.5 [3383.8 to 4870.2] | 3584.8 [2750.7 to 4672.0]
  rSBA-MenC | 13823.5 [10839.7 to 17628.7] | 3444.3 [1998.5 to 5936.0]
  rSBA-MenW-135 | 23431.0 [17351.4 to 31640.7] | 5792.6 [3585.9 to 9357.4]
  rSBA-MenY | 8958.4 [7601.6 to 10557.5] | 5137.8 [3528.2 to 7481.6]

13. Secondary Outcome: Booster Phase: Percentage of Participants With rSBA Booster Response at 1 Month After Booster Vaccination
Description: Serogroups included MenA, MenC, MenW-135 and MenY. rSBA booster vaccine responses for serogroups A, C, W-135 and Y defined as: for initially seronegative participants (pre-vaccination titer below the cut-off of 1:8) had rSBA antibody titers >= 1:32, 1 month after vaccination, and for initially seropositive participants (pre-vaccination titer >= 1:8) had rSBA antibody titers at least 4 times the pre-vaccination antibody titers, 1 month after vaccination. Data reported below is including both seropositive and seronegative participants.
Time Frame: 1 month after booster vaccination
Population: All eligible participants: received primary vaccination in study 107386[NCT00356369] and booster dose in study MENACWY-099;assay results available for antibodies against at least 1 study vaccine antigen component in blood sample taken 1 month post vaccination. N=participants evaluable for measure, n=participants analyzed for specified serogroups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 155 | 52
percentage of participants
  rSBA-MenA | 87.7 [81.5 to 92.5] | 88.5 [76.6 to 95.6]
  rSBA-MenC: number analyzed (Participants) | 154 | 52
  rSBA-MenC | 90.9 [85.2 to 94.9] | 75.0 [61.1 to 86.0]
  rSBA-MenW-135: number analyzed (Participants) | 154 | 52
  rSBA-MenW-135 | 94.2 [89.2 to 97.3] | 96.2 [86.8 to 99.5]
  rSBA-MenY: number analyzed (Participants) | 154 | 52
  rSBA-MenY | 83.8 [77.0 to 89.2] | 92.3 [81.5 to 97.9]

14. Secondary Outcome: Booster Phase: Percentage of Participants With Antibodies Against-Tetanus Toxoid (Anti-TT) Concentrations >=0.1 International Units Per Millilitre (IU/mL), >=1.0 IU/mL at 1 Month After Booster Vaccination
Description: Tetanus toxoid (TT) was used as carrier in tetravalent meningococcal ACWY conjugate vaccine. Percentage of participants with anti-TT concentration >=0.1 IU/mL, >=1.0 IU/mL were summarized.
Time Frame: 1 month after booster vaccination
Population: All eligible participants who received primary vaccination in study107386 [NCT00356369], received booster dose of vaccine in study MENACWY-099; for whom assay results are available for antibodies against at least 1 study vaccine antigen component for blood sample taken 1 month after vaccination. N=participants evaluable for this measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 155 | 52
percentage of participants
  Anti-TT >=0.1 IU/mL | 99.4 [96.5 to 100.0] | 98.1 [89.7 to 100.0]
  Anti-TT >=1.0 IU/mL | 94.8 [90.1 to 97.7] | 88.5 [76.6 to 95.6]

15. Secondary Outcome: Booster Phase: Geometric Mean Concentrations (GMCs) of Antibodies Against-Tetanus Toxoid (Anti-TT) at 1 Month After Booster Vaccination
Description: TT was used as carrier in tetravalent meningococcal ACWY conjugate vaccine. Percentage of participants with anti-TT concentration >=0.1 IU/mL, >=1.0 IU/mL were summarized.
Time Frame: 1 month after booster vaccination
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 155 | 52
IU/mL | 7.163 [5.958 to 8.613] | 7.650 [4.888 to 11.973]

16. Secondary Outcome: Booster Phase: Percentage of Participants With Solicited Local and General Adverse Events up to 4 Days Post Booster Vaccination
Description: Solicited local events:1)pain(Grade [G] : 0=none,1=mild,neither interfered nor prevented normal activities,2=moderate, painful when limb moved; interfered with normal activities,3=severe, significant pain at rest,prevented normal activities),2)redness, and 3)swelling (record greatest surface diameter in millimetre[mm] as 0 to less than or equal to[<=]20 mm, greater than[>]20 to <=50 mm,>50 mm). If to resolve any event medical advice taken, results reported as Medical Advice. Solicited general events: 1) fatigue, 2) gastrointestinal(GI) events(nausea, vomiting, diarrhea and/or abdominal pain,3) headache(G : 0=normal, 1=mild, easily tolerated,2=moderate, interfered with normal activity,3=severe, prevented normal activity), and 4)fever (G: 0=less than[<] 37.5 degree Celsius[°C], 1= 37.5 degree C to 38.0degree C, 2= 38.1 degreeC to 39.0 degree C,3 =>39.0 degree C). 'Related'=relationship to study vaccine assessed by investigator.Medical advice=medical advice received to resolve any event.
Time Frame: Up to 4 days post booster vaccination
Population: All eligible participants who received primary vaccination in study 107386 [NCT00356369] and received booster dose of vaccine in study MENACWY-099. "n" participants analyzed for specified categories.
Measure: Number; unit: percentage of participants
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 164 | 56
percentage of participants
  All pain: number analyzed (Participants) | 159 | 53
  All pain | 27.0 | 26.4
  Pain: Grade 1: number analyzed (Participants) | 159 | 53
  Pain: Grade 1 | 20.8 | 24.5
  Pain: Grade 2: number analyzed (Participants) | 159 | 53
  Pain: Grade 2 | 5.7 | 1.9
  Severe pain: Grade 3: number analyzed (Participants) | 159 | 53
  Severe pain: Grade 3 | 0.6 | 0.0
  Pain: Medical advice: number analyzed (Participants) | 159 | 53
  Pain: Medical advice | 0.0 | 0.0
  All redness: number analyzed (Participants) | 159 | 53
  All redness | 5.7 | 3.8
  Redness: 0 to <=20 mm: number analyzed (Participants) | 159 | 53
  Redness: 0 to <=20 mm | 5.7 | 3.8
  Redness: >20 to <=50 mm: number analyzed (Participants) | 159 | 53
  Redness: >20 to <=50 mm | 0.0 | 0.0
  Redness: >50 mm: number analyzed (Participants) | 159 | 53
  Redness: >50 mm | 0.0 | 0.0
  Redness: Medical advice: number analyzed (Participants) | 159 | 53
  Redness: Medical advice | 0.0 | 0.0
  All swelling: number analyzed (Participants) | 159 | 53
  All swelling | 3.8 | 5.7
  Swelling: 0 to <=20 mm: number analyzed (Participants) | 159 | 53
  Swelling: 0 to <=20 mm | 3.8 | 5.7
  Swelling: >20 to <=50 mm: number analyzed (Participants) | 159 | 53
  Swelling: >20 to <=50 mm | 0.0 | 0.0
  Swelling: >50 mm: number analyzed (Participants) | 159 | 53
  Swelling: >50 mm | 0.0 | 0.0
  Swelling: Medical advice: number analyzed (Participants) | 159 | 53
  Swelling: Medical advice | 0.0 | 0.0
  All fatigue: number analyzed (Participants) | 159 | 53
  All fatigue | 14.5 | 15.1
  Fatigue: Grade 1: number analyzed (Participants) | 159 | 53
  Fatigue: Grade 1 | 10.7 | 15.1
  Fatigue: Grade 2: number analyzed (Participants) | 159 | 53
  Fatigue: Grade 2 | 3.1 | 0.0
  Fatigue: Grade 3: number analyzed (Participants) | 159 | 53
  Fatigue: Grade 3 | 0.6 | 0.0
  Fatigue: Related fatigue: number analyzed (Participants) | 159 | 53
  Fatigue: Related fatigue | 12.6 | 15.1
  Fatigue: Grade 3 Related: number analyzed (Participants) | 159 | 53
  Fatigue: Grade 3 Related | 0.6 | 0.0
  Fatigue: Medical advice: number analyzed (Participants) | 159 | 53
  Fatigue: Medical advice | 0.0 | 0.0
  All fever: number analyzed (Participants) | 159 | 53
  All fever | 6.9 | 5.7
  Fever: Grade 1: number analyzed (Participants) | 159 | 53
  Fever: Grade 1 | 6.3 | 5.7
  Fever: Grade 2: number analyzed (Participants) | 159 | 53
  Fever: Grade 2 | 0.6 | 0.0
  Fever: Grade 3: number analyzed (Participants) | 159 | 53
  Fever: Grade 3 | 0.0 | 0.0
  Fever: Related: number analyzed (Participants) | 159 | 53
  Fever: Related | 6.9 | 5.7
  Fever: Grade 3 related: number analyzed (Participants) | 159 | 53
  Fever: Grade 3 related | 0.0 | 0.0
  Fever: Medical advice: number analyzed (Participants) | 159 | 53
  Fever: Medical advice | 0.0 | 0.0
  All GI: number analyzed (Participants) | 159 | 53
  All GI | 4.4 | 1.9
  GI: Grade 1: number analyzed (Participants) | 159 | 53
  GI: Grade 1 | 3.8 | 1.9
  GI: Grade 2: number analyzed (Participants) | 159 | 53
  GI: Grade 2 | 0.0 | 0.0
  GI: Grade 3: number analyzed (Participants) | 159 | 53
  GI: Grade 3 | 0.6 | 0.0
  GI: Related: number analyzed (Participants) | 159 | 53
  GI: Related | 3.8 | 1.9
  GI: Grade 3 related: number analyzed (Participants) | 159 | 53
  GI: Grade 3 related | 0.6 | 0.0
  GI:Medical advice: number analyzed (Participants) | 159 | 53
  GI:Medical advice | 0.0 | 0.0
  All headache: number analyzed (Participants) | 159 | 53
  All headache | 15.7 | 9.4
  Headache: Grade 1: number analyzed (Participants) | 159 | 53
  Headache: Grade 1 | 12.6 | 9.4
  Headache: Grade 2: number analyzed (Participants) | 159 | 53
  Headache: Grade 2 | 1.9 | 0.0
  Headache: Grade 3: number analyzed (Participants) | 159 | 53
  Headache: Grade 3 | 1.3 | 0.0
  Headache: Related: number analyzed (Participants) | 159 | 53
  Headache: Related | 13.8 | 9.4
  Headache: Grade 3 related: number analyzed (Participants) | 159 | 53
  Headache: Grade 3 related | 1.3 | 0.0
  Headache: Medical advice: number analyzed (Participants) | 159 | 53
  Headache: Medical advice | 0.0 | 0.0

17. Secondary Outcome: Booster Phase: Percentage of Participants With Unsolicited Adverse Events (AEs) up to 31 Days Post Booster Vaccination
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An unsolicited AE covers any untoward medical occurrence in a clinical investigation participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Up to 31 days post booster vaccination
Population: All eligible participants who received primary vaccination in study 107386 [NCT00356369] and received booster dose of vaccine in study MENACWY-099.
Measure: Number; unit: percentage of participants
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 164 | 56
percentage of participants | 9.1 | 3.6

18. Secondary Outcome: Booster Phase: Percentage of Participants With Serious Adverse Events (SAEs) From Booster Vaccination up to End of Study (6 Months Post Booster Vaccination)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Up to 6 months post booster vaccination
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 164 | 56
percentage of participants | 0 | 0

19. Secondary Outcome: Booster Phase: Percentage of Participants With New Onset Chronic Illness From Booster Vaccination up to End of Study (6 Months Post Booster Vaccination)
Description: New onset chronic illness included autoimmune disorders, asthma, type I diabetes, and allergies.
Time Frame: Up to 6 months post booster vaccination
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 164 | 56
percentage of participants | 0 | 0

20. Secondary Outcome: Booster Phase: Percentage of Participants With Guillain-Barre Syndrome (GBS) From Booster Vaccination up to End of Study (6 Months Post Booster Vaccination)
Description: Guillain-Barre syndrome (GBS) is a rare neurological disorder in which the body's immune system mistakenly attacks part of its peripheral nervous system-the network of nerves located outside of the brain and spinal cord. GBS can range from a very mild case with brief weakness to nearly devastating paralysis, leaving the person unable to breathe independently.
Time Frame: Up to 6 months post booster vaccination
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 164 | 56
percentage of participants | 0 | 0

21. Secondary Outcome: Booster Phase: Percentage of Participants With Meningococcal Disease From Booster Vaccination up to End of Study (6 Months Post Booster Vaccination)
Description: Meningococcal disease describes infections caused by the bacterium Neisseria meningitidis (also termed meningococcus). It causes two life threatening diseases: meningococcal meningitis and fulminant meningococcemia which often occur together. Meningococcal meningitis is defined as an inflammatory response to bacterial infection of leptomeninges (pia-arachnoid) and the sub-arachnoid space. Meningococcal meningococcemia is meningococcal septicemia when the bacteria circulate and multiply in blood and involve multiple organs. It can cause multi-organ failure and severe disability or death.
Time Frame: Up to 6 months post booster vaccination
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 164 | 56
percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: For persistence phase: Through 4 years (7, 8, 9 and 10 years post primary vaccination) Non-SAEs were not collected for persistence phase; Booster phase: up to 6 months after booster vaccination; Local and General reactions: Recorded by participants in e-diary up to 4 days post booster vaccination.
Description: Same event may appear as both AE and SAE. What is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in other, or participant may have experienced both serious and non-serious event. Persistence Phase: included all the participants enrolled in the study MENACWY-099. Booster Phase: all eligible participants who received primary vaccination in study 107386[NCT00356369] and booster vaccine in study MENACWY-099.
Groups:
- Persistence Phase: ACWY-TT Group; Booster Phase: ACWY-TT Group: Persistence phase was followed up by booster phase. Persistence phase: Participants received a single 0.5 mL dose of MenACWY-TT vaccine intramuscularly, as primary vaccination in study 107386 [NCT00356369]. Then, in this study (MENACWY-TT-99), they were evaluated for long-term persistence (of immune response) for 4 years (7, 8, 9 and 10 years post primary vaccination). Booster phase: All eligible participants from persistence phase who provided informed consent to enroll in booster phase, received a single 0.5 mL booster dose of MenACWY-TT vaccine intramuscularly in this study, 10 years post primary vaccination in 107386 [NCT00356369], and were followed up for 6 months after booster vaccination.
- Persistence Phase: MenPS Group; Booster Phase: MenPS Group: Persistence phase was followed up by booster phase. Persistence phase: Participants received a single 0.5 mL dose of Mencevax ACWY vaccine intramuscularly, as primary vaccination in study 107386 [NCT00356369]. Then, in this study (MENACWY-TT-99) they were evaluated for long-term persistence (of immune response) for 4 years (7, 8, 9 and 10 years post primary vaccination). Booster phase: All eligible participants from persistence phase who provided informed consent to enroll in booster phase, received a single 0.5 mL booster dose of MenACWY-TT vaccine intramuscularly in this study, 10 years post primary vaccination, and were followed up for 6 months after booster vaccination.
Arm/Group | Persistence Phase: ACWY-TT Group | Persistence Phase: MenPS Group | Booster Phase: ACWY-TT Group | Booster Phase: MenPS Group
All-Cause Mortality (participants affected / at risk) | 0/235 | 0/76 | 0/164 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/235 | 0/76 | 0/164 | 0/56
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 66/164 | 20/56
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Persistence Phase: ACWY-TT Group (N=0) | Persistence Phase: MenPS Group (N=0) | Booster Phase: ACWY-TT Group (N=164) | Booster Phase: MenPS Group (N=56)
Gastrointestinal (Gastrointestinal disorders) | 0 | 0 | 7 | 1
Fatigue (General disorders) | 0 | 0 | 23 | 8
Influenza like illness (General disorders) | 0 | 0 | 2 | 0
Injection site erythema (redness) (General disorders) | 0 | 0 | 9 | 2
Injection site pain (pain at injection site) (General disorders) | 0 | 0 | 43 | 14
Injection site swelling (swelling) (General disorders) | 0 | 0 | 6 | 3
Nasopharyngitis (Infections and infestations) | 0 | 0 | 3 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 3 | 0
Headache (Nervous system disorders) | 0 | 0 | 25 | 5

LIMITATIONS AND CAVEATS:
Enrollment for this study (MENACWY-TT-99) started at Year 6. However, Study visit for Year 6 was not done because approval was not obtained from the authorities until after the end of the Year 6. Hence, no planned activities were done for Year 6.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-02-29): https://cdn.clinicaltrials.gov/large-docs/40/NCT01934140/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT01934140/SAP_001.pdf